CLINICAL TRIAL: NCT04995432
Title: Non Contrast MRI in Lower Extremity: Role in Varicose Vein , Stasis Ulcer and Obstructive Venous Disease
Brief Title: Non Contrast MRI in Lower Extremity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201901058B0 and 202001213B0
Record Dates: First submitted 2021-08-02; First posted 2021-08-09 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-06

CONDITIONS: Venous Insufficiency of Leg; Venous Leg Ulcer; Venous Occlusion; Contrast Media Reaction
Keywords: MRI, CVS; contrast; reflux; ablation
MeSH Terms: conditions — Varicose Ulcer; Familial cyclic vomiting syndrome; Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
We collected retrospectively the non contrast MRI in chia yi memorial hospital for different venous disease of lower extremity morphology and flow ananlysis were done.

DETAILED DESCRIPTION:
Retrospective, analysis of the venous figure by TRANCE MRI no drug/contrast median usage no radiation toxicity the range from the pelvic to the toe

ELIGIBILITY:
Inclusion Criteria:

* possible venous disease no contraindication for mri

Exclusion Criteria:

* could not tolerate mri packemaker

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: retrospective, patients with leg venous disease
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
image quality | 1 year
  good or artifact

CONTACTS AND LOCATIONS:
Locations (1):
- Yao-Kuang Huang, Chiayi City, Taiwan